CLINICAL TRIAL: NCT00127712
Title: Prevention of Atrial Fibrillation Following Noncardiac Thoracic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other)
Responsible Party: Principal Investigator, James E. Tisdale, Professor and Interim Head, Dept of Pharmacy Practice, Purdue University and Adjunct Professor, School of Medicine, Indiana University, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0407-16
Record Dates: First submitted 2005-08-04; First posted 2005-08-08 (Estimated); Results first posted 2010-03-24 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Atrial Fibrillation
Keywords: amiodarone; atrial fibrillation; surgical procedures, thoracic
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amiodarone (Experimental): Amiodarone 1050 mg via continuous intravenous infusion for 24 hours followed by 400 mg orally twice daily for 6 days
  Interventions: Drug: Amiodarone
- No treatment (No Intervention): Patients in this group receive no intervention

INTERVENTIONS:
Drug: Amiodarone
  Arms: Amiodarone

SUMMARY:
The investigators hypothesize that the medication amiodarone decreases the incidence of atrial fibrillation (AF) following non-cardiac open-chest surgery. Their specific aims are to:

* Determine the effectiveness of amiodarone for the prevention of AF following non-cardiac open-chest surgery;
* Determine the influence of the prevention of AF following non-cardiac thoracic surgery on post-surgical duration of stay in the Intensive Care Unit (ICU); post-surgical duration of stay in a hospital unit that employs cardiac monitoring; and duration of post-surgical hospital stay; and
* Determine the safety of amiodarone for the prevention of AF following non-cardiac open-chest surgery.

DETAILED DESCRIPTION:
Thousands of patients undergo major non-cardiac open-chest surgery in the United States each year. These surgeries most often consist of lung surgery, in which one lobe of the lung is removed (lobectomy) or the entire lung is removed (pneumonectomy).

A major complication of these non-cardiac open-chest surgeries is the occurrence of an irregular heartbeat known as atrial fibrillation (AF), which develops in up to 40% of patients undergoing these procedures. AF is characterized by rapid, irregular, chaotic beating of the two smaller chambers of the heart (the atria), leading to rapid, irregular beating of the two larger chambers (the ventricles). The average time to occurrence of post-surgical AF is 2-3 days following surgery. AF occurring following major non-cardiac open-chest surgery can result in extremely rapid heart rates, as fast as 150-200 beats per minute, and may be associated with serious consequences, including severely low blood pressure and potentially debilitating stroke. Further, the risk of death following non-cardiac open-chest surgery is significantly higher in patients who develop AF compared with those who do not. Therefore, the occurrence of this irregular heartbeat following non-cardiac open-chest surgery is associated with severe, potentially life-threatening consequences. Prevention of this irregular heartbeat in these patients may therefore be very important.

Amiodarone is a medication that is known to be effective for prevention and treatment of AF that occurs in patients who have not undergone surgery. In addition, amiodarone has been shown to be effective for prevention of AF following open-chest heart surgery. However, the use of medications for prevention of AF following non-cardiac open-chest surgery has not been well studied, and amiodarone has not been studied in a controlled trial for the prevention of AF in patients undergoing these procedures. In addition, amiodarone is associated with side effects, and it is important to determine the safety of this medication when used in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Males or females over the age of 40
* Scheduled to undergo pneumonectomy or lobectomy

Exclusion Criteria:

* History (hx) of atrial fibrillation
* Prior severe side effects from amiodarone
* Elevated liver enzymes >3 times the upper limit of normal (UNL)
* QTc interval > 450 ms
* Receiving class Ia or class III antiarrhythmics

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2004-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Tisdale, PharmD, Principal Investigator — Department of Pharmacy Practice- School of Pharmacy and Pharmacal Sciences- Purdue University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Tisdale JE, Wroblewski HA, Wall DS, Rieger KM, Hammoud ZT, Young JV, Kesler KA. A randomized trial evaluating amiodarone for prevention of atrial fibrillation after pulmonary resection. Ann Thorac Surg. 2009 Sep;88(3):886-93; discussion 894-5. doi: 10.1016/j.athoracsur.2009.04.074. PMID 19699916

RESULTS

PARTICIPANT FLOW:
Groups:
- Amiodarone: Determine if amiodarone is effective for prevention of atrial fibrillation ater pulmonary resection surgery
- Control: Control group
Period: Overall Study
Arm/Group | Amiodarone | Control
Started | 65 | 65
Completed | 60 | 65
Not Completed | 5 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Lack of GI access to continue | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amiodarone | Control | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 39 | 83
  >=65 years | 21 | 26 | 47
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (8) | 63 (9) | 62 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 34 | 65
  Male | 34 | 31 | 65
Region of Enrollment [Number; unit: participants]
  United States | 65 | 65 | 130

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Atrial Fibrillation Requiring Treatment
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Amiodarone | Control
Number analyzed (Participants) | 65 | 65
participants | 9 | 21
Statistical Analysis 1: Comparison: Amiodarone vs Control; Test type: Superiority or Other; p = 0.02, Chi-squared

2. Secondary Outcome: Length of Intensive Care Unit Stay
Time Frame: Duration of hospitalization
Measure: Median (Full Range); unit: Hours
Arm/Group | Amiodarone | Control
Number analyzed (Participants) | 65 | 65
Hours | 46 [0 to 1416] | 84 [0 to 984]
Statistical Analysis 1: Comparison: Amiodarone vs Control; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Incidence of Atrial Fibrillation Lasting Longer Than 30 Seconds
Time Frame: 7 days
Measure: Number; unit: Participants
Arm/Group | Amiodarone | Control
Number analyzed (Participants) | 65 | 65
Participants | 9 | 22
Statistical Analysis 1: Comparison: Amiodarone vs Control; Test type: Superiority or Other; p = 0.001, Chi-squared

4. Secondary Outcome: Length of Hospital Stay
Time Frame: Duration of hospitalization
Measure: Median (Full Range); unit: Days
Arm/Group | Amiodarone | Control
Number analyzed (Participants) | 65 | 65
Days | 7 [3 to 59] | 8 [3 to 41]
Statistical Analysis 1: Comparison: Amiodarone vs Control; Test type: Superiority or Other; p = 0.79, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Amiodarone | Control
Serious Adverse Events (participants affected / at risk) | 2/65 | 1/65
Other Adverse Events (participants affected / at risk) | 21/65 | 22/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amiodarone (N=65) | Control (N=65)
death (General disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amiodarone (N=65) | Control (N=65)
Hypotension (General disorders) | 21 (21) | 22 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No